CLINICAL TRIAL: NCT04106271
Title: The Effectiveness of a Dyadic Pain Management Program for Older People and Informal Caregivers With Chronic Pain: A Pilot Randomized Controlled Trial
Brief Title: Dyadic Pain Management Program for Older Adults and Informal Caregivers With Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSE Mun Yee Mimi, Associate professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: DPMCP
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; dyadic pain management program; older adults; informal caregiver
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): dyadic pain management program will be accessible by the intervention group
  Interventions: Other: dyadic pain management program
- Control group (No Intervention): No intervention for the control group, only one-page simple material related to pain will be provided.

INTERVENTIONS:
Other: dyadic pain management program — a dyadic pain management program for older adults and their informal caregivers is developed as intervention. The program will be conducted at community activity center face-to-face combined with digital-based activities and the program will include 4 sessions, weekly 1 hours. Each session will be classified into three stages, including 10 minutes for watching videos and group discussion, 20 minutes for theoretical knowledge and coping skills and 20 minutes for exercising together. Last 10 minutes of each session is to wrap up and Q & A. There will be a brief introduction of program and self-introduction of participants at the beginning of the first session. One exercise book is given to each pair and researchers have a 4-week follow-up.
  Arms: Experimental group

SUMMARY:
Chronic pain is a common health problem among older adults and their informal caregivers. Chronic pain has negative effects on physical and psychological health status and it is a strong predictor of poor quality of life. In this study, a dyadic face-to-face pain management program will be provided to older adults and informal caregivers to help the dyads equip with pain-related knowledge and pain coping skills. The effectiveness of the dyadic program will be assessed. Participants will be recruited follow snowball sampling and will be randomly allocated to experimental group and control group using 1: 1 radio. The dyadic pain management program will last four weeks, including group discussion, pain-related knowledge and physical exercises. Pain intensity, anxiety, depression, stress, pain self-efficacy and quality of life will be measured in baseline, post-treatment and at one-month follow. Acceptability and satisfaction to the program will be collected.

This study will be held in Caritas District Elderly Centre-Yeun Long (Tin Chak Centre) and Caritas Cheng Shing Fung District Elderly Center (Shamshuipo) in Hong Kong. For sample size, no suitable standard deviation and effect size was found in previous similar study through the literature review, so this study will be a pilot RCT study with a total 60 dyads of sample size. 30 older adults and 30 informal caregivers will be in each group (experimental group and control group). The dyadic pain management program will be held in the community activity center at weekends and will involve three parts: demographic data, outcome measures (baseline, post-treatment and one-month follow-up measures) and pain education.

Potential participants' eligibility will be confirmed by a questionnaire designed according to inclusion criteria and exclusion criteria. An information sheet will be provided to the eligible dyads and informed consent will be signed on the scene. Experimental group will start pain management program when finish the baseline assessment and control group will be given one page of pain management information download from Department of Health. (http://www.elderly.gov.hk/english/common_health_problems/bones_and_joints/index.html). For optimal communication, two WhatsApp groups will be created consisting of all the caregivers in experimental group and control group respectively.

Outcomes will be measured at three times during the whole intervention, T0 baseline prior to intervention, T1 in week four when the experimental group finish all the program and T2 in week eight with one-month follow-up after the program. Dyads' demographic and caregiving-related questions will be completed prior to beginning the program in T0. Pain related situations, anxiety, depression, stress, quality of life, pain self-efficacy will be measured from older adults and informal caregivers at T0, T1, T2, using a same battery of questionnaires. Dyads' acceptability and satisfaction will be administered immediately after the last session. Data will be collected by a research assistant blinded to the dyads' group assignments.

DETAILED DESCRIPTION:
Participants

This study is a dyadic intervention. Target populations are older adults and informal caregivers with chronic pain. A pair of informal caregiver and older adult will be regarded as a dyad. Dyads will be recruited in the community following the snowball sampling, the eligibility will be accessed based on the following details:

Older adults

Inclusion criteria for older adults:

1. Aged 65 or above;
2. Have an informal caregiver willing to participate this program;
3. Can understand Chinese;
4. Have a history of non-cancer pain in past 6 months;
5. Pain score should be at least 2 measured by Numeric Rating Scale, a 11-point numeric scale ;
6. Have behavioral abilities to do a light exercise and stretch program;
7. Able to attend the whole sessions in community activity center.

Exclusion criteria for older adults:

1. Have serious organic disease or malignant tumor;
2. Have a history of consciousness or mental disorder diagnosed by neurologists or psychiatrists;
3. Have a further medical/surgical treatment in two months or have joined in other pain management program.
4. Experience a drug addiction problem

Informal caregivers Inclusion criteria for informal caregivers

1. Aged 18 or above;
2. As an informal caregiver for one older adult;
3. Can understand Chinese;
4. Have a history of non-cancer pain in past 6 months;
5. Pain score should be at least 2 measured by Numeric Rating Scale, a 11-point numeric scale ;
6. Own a smartphone and can assess the internet;
7. Able to attend the whole sessions in community activity center.

Exclusion criteria for informal caregivers

1. Have serious organic disease or malignant tumor;
2. Have a history of consciousness or mental disorder diagnosed by neurologists or psychiatrists;
3. Have a further medical/surgical treatment in two months or have joined in other pain management program.
4. Experience a drug addiction problem

Outcome measures It is a dyadic intervention so outcomes will be measured from older adults and informal caregivers.

Primary outcome The Brief Pain Inventory-Chinese Version It is a tool to evaluate the intensity, site, quality, relief, interference and causes of pain in patients. Four items for the degree of pain severity, one item for the degree of pain relief and seven items for degree of pain interferes will assess, numbering the different pain sites from 0 to 10. For BPI-C, the Cronbach's α for the pain severity and pain interference items are 0.83-0.89 and 0.90-0.91 and has good acceptable test-retest reliability .

Secondary outcomes:

World Health Organization Quality of Life-Brief It is a self-report questionnaire which assesses 4 domains of quality of life, including physical health, psychological health, social relationships, and environment. Participants will express how much they have experienced in the preceding two weeks on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely). Previous studies showed that WHOQOL-BRIF has good internal consistency and validity.

Depression Anxiety Stress Scale It is a self-administered psychological instrument to evaluate the degree of depression, anxiety and stress involving 21 items. Every part has seven items on a 4-point Likert scale ranging from 0 to 3. The instrument was used in previous studies and had good internal consistency and validity.

Pain Self-efficacy Questionnaire It is a tool to measure the self-efficacy in coping with daily activities with pain . A Chinese version of the PSEQ will be used in this study. Participants will express participants' confidence in performing ten activities experiencing pain on a 7-point Likert scale ranging from 0 (not at all confident) to 6 (completely cinfident). Previous studies illustrated the test-rest reliability coefficient of PSEQ was 0.75 and internal consistency, Cronbach's alpha was 0.95, which was reliable .

Satisfaction and acceptability Participants' satisfaction and acceptability of the dyadic intervention will be assessed at the end of the grogram. Some open-ended questions will be asked, including "What topics, content, or concepts could have been covered in more/less detail?" "As a result of participating in dyadic pain management intervention, did you make some positive changes in your life?" "Would you feel the group discussions interesting and informative? Did the activities and exercises relieve your pain symptom?" These questions were used in previous studies to evaluate the satisfaction and acceptability of intervention program.

ELIGIBILITY:
Inclusion Criteria:

For Older adults:

1. Aged 65 or above;
2. Have an informal caregiver willing to participate this program;
3. Can understand Chinese;
4. Have a history of non-cancer pain in past 6 months;
5. Pain score should be at least 2 measured by Numeric Rating Scale, a 11-point numeric scale;
6. Have behavioral abilities to do a light exercise and stretch program;
7. Able to attend the whole sessions in community activity center.

For Informal caregivers:

1. Aged 18 or above;
2. As an informal caregiver for one older adult;
3. Can understand Chinese;
4. Have a history of non-cancer pain in past 6 months;
5. Pain score should be at least 2 measured by Numeric Rating Scale, a 11-point numeric scale;
6. Own a smartphone and can assess the internet;
7. Able to attend the whole sessions in community activity center.

Exclusion Criteria:

For Older adults:

1. Have serious organic disease or malignant tumor;
2. Have a history of consciousness or mental disorder diagnosed by neurologists or psychiatrists;
3. Have a further medical/surgical treatment in two months or have joined in other pain management program.
4. Experience a drug addiction problem.

For Informal caregivers:

1. Have serious organic disease or malignant tumor;
2. Have a history of consciousness or mental disorder diagnosed by neurologists or psychiatrists;
3. Have a further medical/surgical treatment in two months or have joined in other pain management program.
4. Experience a drug addiction problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2022-06-28 (Estimated); Study Completion 2022-06-28 (Estimated)

PRIMARY OUTCOMES:
Pain intensity and pain interference | Baseline, Week 4, one-month after intervention
  Changes from baseline to Week 4 and one-month after the intervention in pain intensity and pain interference using Brief Pain Inventory

SECONDARY OUTCOMES:
Depression, Anxiety and Stress | Baseline, Week 4, one-month after intervention
  Changes from baseline to Week 4 and one-month after the intervention in depression, anxiety and stress using Depression Anxiety Stress Scale - 21 Scale (DASS-21#. The DASS-21 is a set of three self-reported scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items and divided into subscales. The score of each item ranges feom 0 to 3 (o = do not apply to me at all, 3 = applied to me very much or most of the time). Total score is multiplied by 2 of the sum of each subscales. Higher score indicates the greater degree of the symptom.
Pain self-efficacy | Baseline, Week 4, one-month after intervention
  Changes from baseline to Week 4 and one-month after the intervention in pain self-efficacy using Pain Self-Efficacy Questionnaire (PSEQ). PSEQ is a 10-item questionnaire assessing the confidence people with ongoing pain have in performing activities while in pain. Score of each item ranges from 0 to 6 (0 = not at all confident, 6 = completely confident). A total score is calculated by adding the scores for each item which ranging from 0 to 60. Higher scores reflect stronger self-efficacy beliefs.
World Health Organization Quality of Life-Brief | Baseline, Week 4, one-month after intervention
  Changes from baseline to Week 4 and one-month after the intervention in quality of life using World Health Organization Quality of Life-Brief. It is a self-report questionnaire which assesses 4 domains of quality of life, including physical health, psychological health, social relationships, and environment. Participants will express how much they have experienced in the preceding two weeks on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely).
Participant's Satisfaction and acceptability to the program | week 4
  Participants satisfaction and acceptability to the online pain education program will be assessed at post-treatment by several questions, including "do you think this online pain education program useful?" "does it worth your time following the program?" "would you feel confident to recommend this program to others?" Participants are required to answer the questions by "Yes" or "No". Open-ended question "what are the advantages and disadvantages of the program?" will also be asked. These questions have in the previous studies to assess the acceptability and satisfaction to the internet-delivered program.

CONTACTS AND LOCATIONS:
Overall Officials: Tse Tse, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No